CLINICAL TRIAL: NCT02359864
Title: Phase I Feasibility Study of Low Dose Whole Brain Irradiation in the Treatment of Alzheimer's Disease
Brief Title: Study of Low Dose Whole Brain Irradiation in the Treatment of Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing and budget limitations. Administrative decision to halt enrollment due to coronavirus-19 (COVID) pandemic
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, James Fontanesi, MD, Staff physician, Radiation Oncology, Corewell Health East
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-088; 2017-471
Record Dates: First submitted 2015-01-30; First posted 2015-02-10 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer's Disease
Keywords: radiation treatment
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single group pilot study of radiation treatment. The two arms are sequential dose increase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort One (Experimental): An initial 15 patients will be enrolled in the first treatment scheme (5 daily fractions of 2 Gy) and will be followed for 12 months after completion of treatment to assess safety and any toxicity/adverse events associated with treatment. 15 patients will be enrolled and each will be followed for 12 months to assess safety and toxicity/adverse events.
  Interventions: Radiation: 5 daily fractions of 2 Gy
- Cohort Two (Experimental): The second treatment arm will not be used until the last patient in the first dose arm has completed all follow up. At that point patients
  #16-30 will be enrolled in the second dose arm (10 daily fractions of 2 Gy). 15 patients will be enrolled and each will be followed for 12 months to assess safety and toxicity/adverse events.
  Interventions: Radiation: 10 daily fractions of 2 Gy

INTERVENTIONS:
Radiation: 5 daily fractions of 2 Gy — Whole Brain Irradiation to treat Alzheimer's Disease
  Arms: Cohort One
Radiation: 10 daily fractions of 2 Gy — Whole Brain Irradiation to treat Alzheimer's Disease
  Arms: Cohort Two

SUMMARY:
This study is designed to assess the safety and toxicity/adverse events associated with the use of low dose fractionated whole brain irradiation in those patients who have been diagnosed with probable Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria. As a secondary goal it will establish whether or not the intervention with low dose whole brain irradiation might change the recognized progression of Alzheimer's Disease. The investigators will also collect information from the florbetaben F 18 Injection (AMYVID®) positron emission tomography (PET) Scans to determine if there is any correlation between neurocognitive/quality of life scores and changes in amyloid plaque size, number and location.

DETAILED DESCRIPTION:
An initial 15 patients will be enrolled in the first treatment scheme (5 daily fractions of 2 Gy) and will be followed for 12 months after completion of treatment to assess safety and any toxicity/adverse events associated with treatment. In Arm 1 the 15 study participants will be enrolled in total at Botsford Radiation Oncology Center and William Beaumont Hospital (Royal Oak Campus). Once a total combined 15 patients are entered this Arm will be closed.

The second treatment arm will not be used until the last patient in the first dose arm has completed all follow up. At that point patients #16-30 will be enrolled in the second dose arm (10 daily fractions of 2 Gy). In Arm 2 the 15 study participants will be enrolled in total at both Botsford Hospital Radiation Oncology Center and William Beaumont Hospital (Royal Oak Campus). Once a total combined 15 patients are entered this Arm will be closed.

A total of 30 patients will be enrolled and each will be followed for 12 months to assess safety and toxicity/adverse events.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Eligibility (All responses must be YES)

Inclusion Criteria:

Patients must meet all eligibility criteria to be included in the study:

1. Must be 55 years of age or older
2. Patient must meet NINCDS-ADRDA criteria for Alzheimer's Disease
3. Patient must be able to complete Mini-Mental Examination (MMSE) and Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) questionnaire Score Sheets
4. Patient has a Rosen Modified Hachinski Ischemic Score of less than or equal to 4
5. Patient has a MMSE score of between 10-20
6. Patient has estimated survival of greater than 12 months
7. Patient or legally authorized representative must be able to give consent

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. The patient has a history of cancer except non-melanoma skin cancer
2. Patient is taking anti-epileptic medication.
3. Dermatological skin disease of the scalp
4. Patient taking Alzheimer medication within the last 3 months, i.e. Exelon, Aricept, Namenda, Reminyl or Ebixa.
5. Current presence of a clinically significant major psychiatric disorder (e.g. major depressive disorder, bipolar disorder, schizophrenia, etc., according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV))
6. Patient currently participating in another Clinical Trial.
7. Patient and legally authorized representative unable to give informed consent
8. Patient with history of focal neurological deficits (with the exception of vibratory peripheral neuropathy)
9. Non-Alzheimer dementia
10. Patient has previous history of central nervous system radiation
11. Patient has evidence of substance abuse (alcohol / or other drugs of dependence) during previous 12 months
12. History of subdural hygroma / subdural hematoma
13. History of cerebral infection / hemorrhage.
14. History that the patient is immunocompromised
15. History of seizure activity
16. History of hydrocephalus

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fontanesi, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Beaumont Health, Farmington Hills, Michigan
  - Beaumont Health, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort Two: The second treatment arm will not be used until the last patient in the first dose arm has completed all follow up. At that point patients
  #16-30 will be enrolled in the second dose arm (10 daily fractions of 2 Gy). 15 patients will be enrolled and each will be followed for 12 months to assess safety and toxicity/adverse events.
  10 daily fractions of 2 Gy: Whole Brain Irradiation to treat Alzheimer's Disease
Period: Overall Study
Arm/Group | Cohort One | Cohort Two
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No enrollment in Cohort 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort One | Cohort Two | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 74.5 [65 to 84] |  | 74.5 [65 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Common Terminology Toxicity Criteria for Adverse Events (CTCAE) Version 5.0 - 6 Weeks
Description: To assess a change from baseline in adverse conditions, utilizing Common Terminology Toxicity Criteria (Version 5.0) assessing skin, eyes, ears, and central nervous system at 6 weeks post-treatment. Each condition/event will be given a score based on severity . The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each adverse event (AE): (Grade 1=1 point, Grade 2=2 points, Grade 3=3 points, Grade 4=4 points. Grade 5=5 points) and event scores added to produce a total patient score. Minimum score is zero, which represents no adverse events. Maximum score is 72. A higher score means a worse outcome. The total patient score at baseline subtracted from the total score at 6 weeks is reported. A positive number indicates an increase in adverse conditions, while a negative number indicates decreased adverse conditions.
Time Frame: Baseline to 6 weeks post-treatment
Population: No patients were enrolled in Cohort Two
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
units on a scale | 2 [1 to 3] |

2. Primary Outcome: Common Terminology Toxicity Criteria (CTCAE) Version 5.0 - 3 Months
Description: To assess a change from baseline in adverse conditions, utilizing Common Terminology Toxicity Criteria (Version 5.0) assessing skin, eyes, ears, and central nervous system at 3 months post-treatment. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE: (Grade 1=1 point, Grade 2=2 points, Grade 3=3 points, Grade 4=4 points. Grade 5=5 points) and event scores added to produce a total patient score. Minimum score is zero, which represents no adverse events. Maximum score is 72. A higher score means a worse outcome. The total patient score at baseline subtracted from the total score at 3 months is reported. A positive number indicates an increase in adverse conditions, while a negative number indicates decreased adverse conditions.
Time Frame: Baseline 3 months post-treatment
Population: No patients were enrolled in Cohort Two
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
units on a scale | 1.5 [0 to 3] |

3. Primary Outcome: Common Terminology Toxicity Criteria (Version 5.0) - 6 Months
Description: To assess a change from baseline in adverse conditions, utilizing Common Terminology Toxicity Criteria (Version 5.0) assessing skin, eyes, ears, and central nervous system at 6 months post-treatment. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE: (Grade 1=1 point, Grade 2=2 points, Grade 3=3 points, Grade 4=4 points. Grade 5=5 points) and event scores added to produce a total patient score. Minimum score is zero, which represents no adverse events. Maximum score is 72. A higher score means a worse outcome. The total patient score at baseline subtracted from the total score at 6 months is reported. A positive number indicates an increase in adverse conditions, while a negative number indicates decreased adverse conditions.
Time Frame: 6 months post-treatment
Population: Due to patient withdrawal, only 1 patient in Cohort 1 had 6 month data. No patients enrolled in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | 0 [0 to 0] |

4. Primary Outcome: Common Terminology Toxicity Criteria (Version 5.0) - 12 Months
Description: To assess a change from baseline in adverse conditions, utilizing Common Terminology Toxicity Criteria (Version 5.0) assessing skin, eyes, ears, and central nervous system at 12 months post-treatment. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE: (Grade 1=1 point, Grade 2=2 points, Grade 3=3 points, Grade 4=4 points. Grade 5=5 points) and event scores added to produce a total patient score. Minimum score is zero, which represents no adverse events. Maximum score is 72. A higher score means a worse outcome. The total patient score at baseline subtracted from the total score at 12 months is reported. A positive number indicates an increase in adverse conditions, while a negative number indicates decreased adverse conditions.
Time Frame: Baseline to12 months post-treatment
Population: Due to patient withdrawal, only 1 patient with data at 12 months in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | 0 [0 to 0] |

5. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change in "Positive" or "Negative" Determination
Description: The number of patients with a change in amyloid plaque burden on AMYVID PET imaging from baseline to 4 month post-treatment scans, based on an overall "positive" or "negative" determination using Eli-Lilly AMYVID criteria. A positive scan indicates moderate to frequent amyloid neuritic plaques. A negative scan indicates sparse to no neuritic plaques.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
Participants | 0 |

6. Secondary Outcome: Neurocognitive Function - MMSE (Mini Mental Status Exam) 6 Weeks Change From Baseline
Description: Change at 6 weeks post-treatment from the pretreatment neurocognitive evaluation utilizing the Mini Mental Status Exam (MMSE) tool; a 30-point questionnaire for assessing cognitive function. Minimum value 0, maximum value 30. Higher score means better outcome. Pretreatment total score subtracted from 6-week total score will be reported.
Time Frame: Baseline to 6 weeks post-treatment
Population: No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
units on a scale | 1 [0 to 2] |

7. Secondary Outcome: Neurocognitive Function - MMSE (Mini Mental Status Exam) 3 Months Change From Baseline
Description: Change at 3 months post-treatment from the pretreatment neurocognitive evaluation utilizing the Mini Mental Status Exam (MMSE) tool; a 30-point questionnaire for assessing cognitive function. Minimum value 0, maximum value 30. Higher score means better outcome. Pretreatment total score subtracted from 3-month total score will be reported.
Time Frame: Baseline to 3 months post-treatment
Population: 1 patient in Cohort 1 did not complete 3 month MMSE. No enrollment in Cohort 2.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | -7 [-7 to -7] |

8. Secondary Outcome: Neurocognitive Function - MMSE (Mini Mental Status Exam) 6 Months Change From Baseline
Description: Change at 6 months post-treatment from the pretreatment neurocognitive evaluation utilizing the Mini Mental Status Exam (MMSE) tool; a 30-point questionnaire for assessing cognitive function. Minimum value 0, maximum value 30. Higher score means better outcome. Pretreatment total score subtracted from 6-month total score will be reported.
Time Frame: Baseline to 6 months post-treatment
Population: Due to patient withdrawal, MMSE data for only 1 patient in Cohort 1 available. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | 1 [1 to 1] |

9. Secondary Outcome: Neurocognitive Function - MMSE (Mini Mental Status Exam) 12 Months Change From Baseline
Description: Change at 12 months post-treatment from the pretreatment neurocognitive evaluation utilizing the Mini Mental Status Exam (MMSE) tool; a 30-point questionnaire for assessing cognitive function. Minimum value 0, maximum value 30. Higher score means better outcome. Pretreatment total score subtracted from 12-month total score will be reported.
Time Frame: Baseline to 12 months post-treatment
Population: No MMSE data for any patient in Cohort 1 available at 12 months. No enrollment in Cohort Two
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Neurocognitive Function - ADAS-Cog - 6 Weeks Change From Baseline
Description: Change at 6 weeks post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Disease Assessment Scale Cognitive Scales (ADAS-Cog), an 11 part questionnaire that provides a weighted score of cognitive function. Minimum score 0, maximum score 70, with higher score indicating worse outcome. Pretreatment total score subtracted from 6-week total score will be reported. Negative numbers indicate an improvement in cognition. Positive numbers indicate a worsening cognition.
Time Frame: Baseline to 6 weeks post-treatment
Population: Data unavailable to any patient in Cohort 1. No patients were enrolled in Cohort 2.
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Neurocognitive Function - ADAS-Cog - 3 Months Change From Baseline
Description: Change at 3 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Disease Assessment Scale Cognitive Scales (ADAS-Cog), an 11 part questionnaire that provides a weighted score of cognitive function. Minimum score 0, maximum score 70, with higher score indicating worse outcome. Pretreatment total score subtracted from 3-month total score will be reported. Negative numbers indicate an improvement in cognition. Positive numbers indicate a worsening cognition.
Time Frame: Baseline to 3 months post-treatment
Population: Data available for 1 patient in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | -14 [-14 to -14] |

12. Secondary Outcome: Neurocognitive Function - ADAS-Cog - 6 Months Change From Baseline
Description: Change at 6 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Disease Assessment Scale Cognitive Scales (ADAS-Cog), an 11 part questionnaire that provides a weighted score of cognitive function. Minimum score 0, maximum score 70, with higher score indicating worse outcome. Pretreatment total score subtracted from 6-month total score will be reported. Negative numbers indicate an improvement in cognition. Positive numbers indicate a worsening cognition.
Time Frame: Baseline to 6 months post-treatment
Population: No data available for patients in Cohort 1. No enrollment in Cohort 2
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Neurocognitive Function - ADAS-Cog - 12 Months Change From Baseline
Description: Change at 12 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Disease Assessment Scale Cognitive Scales (ADAS-Cog), an 11 part questionnaire that provides a weighted score of cognitive function. Minimum score 0, maximum score 70, with higher score indicating worse outcome. Pretreatment total score subtracted from 12-month total score will be reported. Negative numbers indicate an improvement in cognition. Positive numbers indicate a worsening cognition.
Time Frame: Baseline to 12 months post-treatment
Population: No data available for patients in Cohort 1. No enrollment in Cohort 2
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Neurocognitive Function - QOL-AD - 6 Weeks Change From Baseline
Description: Change at 6 weeks post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Quality of Life Questionnaire (QOL-AD) tool; a 13 item assessment with each question scored on a 4 point scale where 1=poor quality of life and 4=excellent quality of life. A cumulative score from all items will be collected (min 13 indicates poor QOL, max 52 indicates excellent QOL) and pretreatment score subtracted from 6-week score. A negative number indicates a decreased quality of life. A positive number indicates an improved quality of life
Time Frame: Baseline to 6 weeks post-treatment
Population: No patients enrolled in Cohort 2.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
units on a scale | 1.5 [-5 to 8] |

15. Secondary Outcome: Neurocognitive Function - QOL-AD - 3 Months Change From Baseline
Description: Change at 3 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Quality of Life Questionaire (QOL-AD) tool; a 13 item assessment with each question scored on a 4 point scale where 1=poor quality of life and 4=excellent quality of life. A cumulative score from all items will be collected (min 13 indicates poor QOL, max 52 indicates excellent QOL) and pretreatment score subtracted from 3-month score. A negative number indicates a decreased quality of life. A positive number indicates an improved quality of life.
Time Frame: Baseline to 3 months post-treatment
Population: Data available for only one patient in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | -3 [-3 to -3] |

16. Secondary Outcome: Neurocognitive Function - QOL-AD - 6 Months Change From Baseline
Description: Change at 6 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Quality of Life Questionaire (QOL-AD) tool; a 13 item assessment with each question scored on a 4 point scale where 1=poor quality of life and 4=excellent quality of life. A cumulative score from all items will be collected (min 13 indicates poor QOL, max 52 indicates excellent QOL) and and pretreatment score subtracted from 6-month score. A negative number indicates a decreased quality of life. A positive number indicates an improved quality of life.
Time Frame: Baseline to 6 months post-treatment
Population: Data available for only 1 patient in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | -2 [-2 to -2] |

17. Secondary Outcome: Neurocognitive Function - QOL-AD - 12 Months Change From Baseline
Description: Change at 12 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Alzheimer's Quality of Life Questionaire (QOL-AD) tool; a 13 item assessment with each question scored on a 4 point scale where 1=poor quality of life and 4=excellent quality of life. A cumulative score from all items will be collected (min 13 indicates poor QOL, max 52 indicates excellent QOL) and pretreatment score subtracted from 12-month score. A negative number indicates a decreased quality of life. A positive number indicates an improved quality of life.
Time Frame: Baseline to 12 months post-treatment
Population: No data available for any patients in Cohort 1. No enrollment in Cohort 2
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Neurocognitive Function - QUALID- 6 Weeks Change From Baseline
Description: Change at 6 weeks post-treatment from the pretreatment neurocognitive evaluation utilizing The Quality of Life in Late Stage Dementia (QUALID) tool; an 11 item assessment with each question scored on a 5 point scale completed by caregiver, where 5=poor quality of life and 1=excellent quality of life. A cumulative score from all items will be collected (min 11 indicates excellent quality of life, max 55 indicates poor quality of life) and pretreatment score subtracted from 6-week score. A positive number indicates a decreased quality of life. A negative number indicates an improved quality of life.
Time Frame: Baseline to 6 weeks post-treatment
Population: No enrollment in Cohort 2.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
units on a scale | 4 [-3 to 11] |

19. Secondary Outcome: Neurocognitive Function - QUALID- 3 Months Change From Baseline
Description: Change at 3 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Quality of Life in Late Stage Dementia (QUALID) tool; an 11 item assessment with each question scored on a 5 point scale completed by a patient or caregiver, where 5=poor quality of life and 1=excellent quality of life. A cumulative score from all items will be collected (min 11 indicates excellent quality of life, max 55 indicates poor quality of life) and pretreatment score subtracted from 3-month score. A positive number indicates a decreased quality of life. A negative number indicates an improved quality of life.
Time Frame: Baseline to 3 months post-treatment
Population: Data available on 1 patient in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | 3 [3 to 3] |

20. Secondary Outcome: Neurocognitive Function - QUALID- 6 Months Change From Baseline
Description: Change at 6 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Quality of Life in Late Stage Dementia (QUALID) tool; an 11 item assessment with each question scored on a 5 point scale completed by a patient or caregiver, where 5=poor quality of life and 1=excellent quality of life. A cumulative score from all items will be collected (min 11 indicates excellent quality of life, max 55 indicates poor quality of life) and pretreatment score subtracted from 6-month score. A positive number indicates a decreased quality of life. A negative number indicates an improved quality of life.
Time Frame: Baseline to 6 months post-treatment
Population: Data available for only 1 patient in Cohort 1. No enrollment in Cohort 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 1 | 0
units on a scale | 0 [0 to 0] |

21. Secondary Outcome: Neurocognitive Function - QUALID- 12 Months Change From Baseline
Description: Change at 12 months post-treatment from the pretreatment neurocognitive evaluation utilizing The Quality of Life in Late Stage Dementia (QUALID) tool; an 11 item assessment with each question scored on a 5 point scale completed by a patient or caregiver, where 5=poor quality of life and 1=excellent quality of life. A cumulative score from all items will be collected (min 11 indicates excellent quality of life, max 55 indicates poor quality of life) and pretreatment score subtracted from 12-month score. A positive number indicates a decreased quality of life. A negative number indicates an improved quality of life.
Time Frame: 12 months post-treatment
Population: No data available for any patient in Cohort 1. No enrollment in Cohort 2
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Frontal Region of the Brain Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the frontal region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the frontal region, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the frontal region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 22.7 [15.3 to 30.1] |

23. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Parietal Region of the Brain Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the parietal region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the parietal region, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the parietal region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 21.5 [13.8 to 29.2] |

24. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Precuneus Region of the Brain Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the precuneus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the precuneus region, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the precuneus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 24.0 [15.0 to 33.1] |

25. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Anterior Cingulate Gyrus Region of the Brain Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the anterior cingulate gyrus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the anterior cingulate gyrus region, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the anterior cingulate gyrus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 18.7 [17.6 to 19.8] |

26. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Posterior Cingulate Gyrus Region of the Brain Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the posterior cingulate gyrus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the posterior cingulate gyrus region, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the posterior cingulate gyrus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 21.3 [18.7 to 23.9] |

27. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Ratio (SUVr) for Whole Brain Cortex Compared to Cerebellum
Description: SUVr is a measure of the amount of radiotracer activity bound to beta amyloid plaque in an individual region of brain tissue compared to radiotracer activity in the cerebellum, which is rarely involved by neuritic plaques. An elevated ratio >1.10 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the whole brain cortex relative to cerebellum is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number (percentage) indicates an increase in SUVr and more plaque burden in the whole brain cortex relative to cerebellum, while a negative number (percentage) indicates a decrease in SUVr and a reduction in plaque burden in the whole brain cortex relative to cerebellum.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUVr
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUVr | 17.7 [9.3 to 26.2] |

28. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Standard Deviation (SUV StdDev) From Normal Patients in SUVr Values for Frontal Region of the Brain
Description: The metric SUV StdDev from normal utilizes a database of age matched, cognitively normal individuals to compare the SUV ratios for individual regions of the brain. An elevated SUV StdDev > 1.65 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the frontal region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number indicates an increase in SUV StdDev and more plaque burden in the frontal region, while a negative number indicates a decrease in SUV StdDev and a reduction in plaque burden in the frontal region
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUV StdDev
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUV StdDev | 111.3 [90.3 to 132.3] |

29. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Standard Deviation (SUV StdDev) From Normal Patients in SUVr Values for Parietal Region of the Brain
Description: The metric SUV StdDev from normal utilizes a database of age matched, cognitively normal individuals to compare the SUV ratios for individual regions of the brain. An elevated SUV StdDev > 1.65 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the parietal region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number indicates an increase in SUV StdDev and more plaque burden in the parietal region, while a negative number indicates a decrease in SUV StdDev and a reduction in plaque burden in the parietal region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUV StdDev
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUV StdDev | 70.0 [63.2 to 76.7] |

30. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Standard Deviation (SUV StdDev) From Normal Patients in SUVr Values for Precuneus Region of the Brain
Description: The metric SUV StdDev from normal utilizes a database of age matched, cognitively normal individuals to compare the SUV ratios for individual regions of the brain. An elevated SUV StdDev > 1.65 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the precuneus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number indicates an increase in SUV StdDev and more plaque burden in the precuneus region, while a negative number indicates a decrease in SUV StdDev and a reduction in plaque burden in the precuneus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUV StdDev
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUV StdDev | 75.3 [59.4 to 91.2] |

31. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Standard Deviation (SUV StdDev) From Normal Patients in SUVr Values for Anterior Cingulate Gyrus Region of the Brain
Description: The metric SUV StdDev from normal utilizes a database of age matched, cognitively normal individuals to compare the SUV ratios for individual regions of the brain. An elevated SUV StdDev > 1.65 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the anterior cingulate gyrus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number indicates an increase in SUV StdDev and more plaque burden in the anterior cingulate gyrus region, while a negative number indicates a decrease in SUV StdDev and a reduction in plaque burden in the anterior cingulate gyrus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUV StdDev
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUV StdDev | 107.6 [77.5 to 137.6] |

32. Secondary Outcome: Florbetaben F 18 Injection (AMYVID) Positron Emission Tomography (PET) Scan: Change From Baseline to 4 Months in Standardized Uptake Value Standard Deviation (SUV StdDev) From Normal Patients in SUVr Values for Posterior Cingulate Gyrus Region of Brain
Description: The metric SUV StdDev from normal utilizes a database of age matched, cognitively normal individuals to compare the SUV ratios for individual regions of the brain. An elevated SUV StdDev > 1.65 indicates a strong likelihood of significant underlying neuritic plaque burden. The percent change from baseline to 4-month scans in the posterior cingulate gyrus region is reported (percent change is calculated by subtracting baseline value from 4-month value; the result is then divided by the baseline value and multiplied by 100 to give a percentage). A positive number indicates an increase in SUV StdDev and more plaque burden in the posterior cingulate gyrus region, while a negative number indicates a decrease in SUV StdDev and a reduction in plaque burden in the posterior cingulate gyrus region.
Time Frame: Baseline to 4 months post-treatment
Population: No patients enrolled in second arm.
Measure: Mean (Full Range); unit: percent change from baseline SUV StdDev
Arm/Group | Cohort One | Cohort Two
Number analyzed (Participants) | 2 | 0
percent change from baseline SUV StdDev | 149.5 [60.1 to 238.9] |

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over 12 months
Description: No enrollment in Cohort 2
Arm/Group | Cohort One | Cohort Two
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort One (N=2) | Cohort Two (N=0)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited data was collected due to low enrollment influenced by the coronavirus-19 (COVID) pandemic. Some data was missing for some patients due to COVID restrictions on research. One patient withdrew from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02359864/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02359864/ICF_001.pdf